CLINICAL TRIAL: NCT03739905
Title: A Phase IIa Study to Evaluate the Safety and Efficacy of Blood-Brain Barrier (BBB) Opening Using Transcranial MR-Guided Focused Ultrasound in Patients With Alzheimer's Disease
Brief Title: ExAblate Blood-Brain Barrier Opening for Treatment of Alzheimer's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: InSightec (Industry)
Collaborators: Focused Ultrasound Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AL003
Record Dates: First submitted 2018-11-02; First posted 2018-11-14 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Alzheimer Disease
Keywords: Magnetic Resonance guided Focal Ultrasound (MRgFUS); Alzheimer's Disease; ExAblate; Blood Brain Barrier
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Blood Brain Barrier (BBB) Disruption (Experimental): The ExAblate Model 4000 Type 2.0 System
  Interventions: Device: Blood Brain Barrier (BBB) Disruption

INTERVENTIONS:
Device: Blood Brain Barrier (BBB) Disruption — Focal Ultrasound (FUS) involves the application of acoustic energy at low frequencies from over 1000 individual transducers into distinct targets to induce BBB disruption.
  Other Names: ExAblate Neuro

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of the ExAblate® Model 4000 Type 2.0 system as a tool to open the blood-brain barrier (BBB) in patients with probable Alzheimer's Disease (AD).

DETAILED DESCRIPTION:
This study is a prospective, open label, single-arm, non-randomized, phase IIa trial to evaluate the feasibility, safety and efficacy of repeated, BBB opening using the ExAblate® Model Type 2.0 (220 kHz) system. Patients with diagnosis of Probable Alzheimer's Disease may qualify for a clinical trial to have three serial ExAblate BBB disruption procedures in specific areas in the brain.This study will be conducted at a single center in Canada and will enroll up to 30 patients.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female between 50-85 years of age
2. Probable Alzheimer's Disease (AD)
3. If taking concurrent Alzheimer's medication, has been on the medication for at least 2 months with a stable dose for at least 3 months
4. Able to communicate sensations during the ExAblate MRgFUS procedure
5. Ambulatory

Exclusion Criteria:

1. MRI Findings
2. Presence of unknown or MR unsafe devices anywhere in the body
3. Significant cardiac disease or unstable hemodynamic status
4. Relative contraindications to ultrasound contrast agent or PET amyloid tracer
5. History of a bleeding disorder
6. History of liver disease
7. Known cerebral or systemic vasculopathy
8. Significant depression and at potential risk of suicide
9. Any contraindications to MRI scanning
10. Any contraindication to lumbar puncture for collection of cerebral spinal fluid
11. Untreated, uncontrolled sleep apnea
12. History of seizure disorder or epilepsy
13. Severely Impaired renal function
14. Currently in a clinical trial involving an investigational product or non-approved use of a drug or device or in any other type of medical research
15. Chronic pulmonary disorders
16. Positive human immunodeficiency virus (HIV)
17. Known apolipoprotein E allele (ApoE4) homozygosity

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2018-12-06 (Actual); Primary Completion 2025-04-09 (Actual); Study Completion 2025-04-09 (Actual)

PRIMARY OUTCOMES:
Device and procedure related adverse events | 6 months
  Rate of adverse events following each treatment through end of study

SECONDARY OUTCOMES:
BBB Disruption and Closure | Immediately after the end of each ExAblate treatment and 24 hours after each treatment
  MRI images post ExAblate treatment to verify that the BBB was disrupted and subsequently closed
Change in Alzheimer's Disease Assessment Scale-Cognition | Baseline and 6 months
  Mental cognition assessment
Change in Amyloid Tracer uptake | Baseline and Day 8 following the third treatment
  PET scan analysis comparing the Amyloid Tracer uptake on images taken at baseline and after the last treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Neurosurgery, Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Meng Y, Goubran M, Rabin JS, McSweeney M, Ottoy J, Pople CB, Huang Y, Storace A, Ozzoude M, Bethune A, Lam B, Swardfager W, Heyn C, Abrahao A, Davidson B, Hamani C, Aubert I, Zetterberg H, Ashton NJ, Karikari TK, Blennow K, Black SE, Hynynen K, Lipsman N. Blood-brain barrier opening of the default mode network in Alzheimer's disease with magnetic resonance-guided focused ultrasound. Brain. 2023 Mar 1;146(3):865-872. doi: 10.1093/brain/awac459. PMID 36694943
- [Derived] Mathew AS, Gorick CM, Price RJ. Multiple regression analysis of a comprehensive transcriptomic data assembly elucidates mechanically- and biochemically-driven responses to focused ultrasound blood-brain barrier disruption. Theranostics. 2021 Oct 11;11(20):9847-9858. doi: 10.7150/thno.65064. eCollection 2021. PMID 34815790
- [Derived] Meng Y, Pople CB, Suppiah S, Llinas M, Huang Y, Sahgal A, Perry J, Keith J, Davidson B, Hamani C, Amemiya Y, Seth A, Leong H, Heyn CC, Aubert I, Hynynen K, Lipsman N. MR-guided focused ultrasound liquid biopsy enriches circulating biomarkers in patients with brain tumors. Neuro Oncol. 2021 Oct 1;23(10):1789-1797. doi: 10.1093/neuonc/noab057. PMID 33693781